CLINICAL TRIAL: NCT03416244
Title: A Multicenter Open-label Phase II Trial to Evaluate Nivolumab and Ipilimumab for 2nd Line Therapy in Elderly Patients With Advanced Esophageal Squamous Cell Cancer
Acronym: RAMONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-STO-0117; 2017-002056-86 (EudraCT Number); CA209-9DD (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Cancer; Oesophageal Cancer; Oesophageal Cancer Metastatic; Esophageal Cancer Metastatic; Esophageal Cancers NOS; Oesophageal Cancer Nos; GastroEsophageal Cancer; Gastrooesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Nivolumab / Ipilimumab combination treatment (Experimental): Nivolumab 240 mg fixed dose IV every 2 weeks; Additionally, after 7 week safety assessment Ipilimumab 1mg/kg IV every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- B. Nivolumab monotherapy (Experimental): Nivolumab 240 mg fixed dose IV every 2 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg IV fixed dose every two weeks
Drug: Ipilimumab — Ipilimumab 1mg/kg IV every six weeks (starting in week 7 after safety assessment)
  Arms: A: Nivolumab / Ipilimumab combination treatment

SUMMARY:
Cancer - including esophageal squamous cell cancer (ESCC) - is a disease of the elderly but little is known about the biology and progression of cancers in these patients.

While most patients receive chemotherapy and/or chemo-radiation as first treatment, no treatment standard for following treatments has been established so far and there is a clear unmet medical need, especially for elderly patients.

Hence, this study assesses the efficacy and safety of two experimental immunotherapy regimens (Nivolumab monotherapy or Nivolumab/Ipilimumab combination) in elderly patients with advanced esophageal squamous cell cancer.

DETAILED DESCRIPTION:
Cancer - including esophageal squamous cell cancer (ESCC) - is a disease of the elderly, more than 60% of all tumors arise in patients with the age of 65 years or older. In contrast, little is known about the biology and progression of cancers in these patients, since most clinical trials enroll patients with age limits of 70 or 75 years.

While most patients undergo chemotherapy and/or chemo-radiation in first-line, the role of second-line therapy is less well understood. No treatment standard has been established so far and there is a clear unmet medical need. This is particularly true for geriatric patients for whom palliative systemic therapies are especially challenging.

Hence, the primary objective of this trial is to demonstrate a significant survival benefit of two experimental immunotherapy regimens (Nivolumab monotherapy or Nivolumab/Ipilimumab combination) in elderly patients with advanced esophageal squamous cell cancer compared to historical data of standard chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent including participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening Evaluations
2. Age ≥ 65 years at time of study entry
3. Histologically confirmed advanced stage non-resectable esophageal squamous cell carcinoma beyond frontline therapy*:

   * stage 4 OR
   * stage 3 non-responder to radio-chemotherapy OR
   * any relapse after chemo-radiation OR
   * any relapse after surgery if patient is ineligible or intolerant to standard frontline therapies OR refuses other treatment * Frontline therapy is defined as chemotherapy (+/-radiotherapy) (e.g. CROSS, FLOT or similar protocols) OR any palliative systemic chemotherapy
4. Geriatric status: SlowGo or GoGo according to G8 and DAFI assessment (G8 > 14 points or CGA/DAFI 0.2 < 0.35)
5. At least 1 measurable lesion according to RECIST 1.1
6. Karnofsky performance status ≥ 50
7. Sufficient cardiac functional reserve defined as ejection fraction ≥ 50%
8. Adequate blood count, liver-enzymes, and renal function:

   * neutrophil count > 1.5 x 10^6/mL
   * WBC ≥ 3000/μL
   * Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3)
   * hemoglobin ≥ 9 g/dL
   * INR ≤ 1.5 and PTT ≤ 1.5 x ULN during the last 7 days before therapy
   * AST (SGOT)/ALT (SGPT) < 3 x institutional upper limit of normal (5 x lower limit in case of liver metastases)
   * bilirubin < 1.5 x ULN
   * Serum creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula below):

   Female CrCl = (140 - age in years) x weight in kg x 0.85 / 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL
9. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving Nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational products (Nivolumab, Ipilimumab). Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception)
10. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Patients < 65 years of age
2. Frail patients (DAFI score ≥ 0.35)
3. Esophageal adenocarcinomas, neuroendocrine tumors
4. Prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including Ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
5. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer
6. Previous treatment in the present study (does not include screening failure).
7. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

   1. Major surgery ≤ 28 days prior first dose of study treatment
   2. Anticancer treatment during the last 30 days prior to start of Nivolumab monotherapy treatment, including systemic therapy or major surgery [palliative radiotherapy has to be completed at least 2 weeks prior to start of study treatment]
   3. History of interstitial lung disease
   4. Known acute or chronic pancreatitis
   5. Known active HBV, HCV or HIV infection
   6. Active tuberculosis
   7. Any other active infection (viral, fungal or bacterial) requiring systemic therapy
   8. History of allogeneic tissue/solid organ transplant
   9. Diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Nivolumab monotherapy treatment.
   10. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
   11. Live vaccine within 30 days prior to the first dose of Nivolumab monotherapy treatment or during study treatment.
   12. Other clinically significant active malignancy requiring treatment OR less then 5 years disease free interval of another primary malignancy
   13. Clinically significant or symptomatic cardiovascular/cerebrovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before enrollment
   14. History or clinical evidence of CNS metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: i. are asymptomatic AND ii. have no requirement for steroids 6 weeks prior to start of Nivolumab monotherapy treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
8. Medication that is known to interfere with any of the agents applied in the trial
9. Has known hypersensitivity to Nivolumab or Ipilimumab or any of the constituents of the products
10. Any other efficacious cancer treatment except protocol specified treatment at study start
11. Patient has received any other investigational product within 28 days of study entry
12. Patient has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. [Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.]
13. Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessaries (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
14. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
15. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
16. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Overall survival | 36 months
  OS measured from first dose of 2nd line therapy to the date of death

SECONDARY OUTCOMES:
Time to QoL deterioration | 36 months
  Time to QoL deterioration defined as a loss of ≥ 10 points in the EORTC QLQ-C30 compared to base-line
Progression free survival | 36 months
  Time from first dosing date to the date of the first documented tumor progression
Objective Response rate | 36 months
  Proportion of treated subjects with response from baseline
Duration of response | 36 months
  Time from first confirmed response to the date of the documented progressive disease or death
Duration of treatment | 36 months
  Time from date of first dose of Nivolumab monotherapy until permanent discontinuation of either NIVO mono therapy or NIVO/IPI combination treatment.
Cumulative dose intensity | 36 months
  Cumulative dose for each IMP
Quality of Life C30 | 36 months
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire (30 items) Version 3.0. The QLQ-C30 is composed of multi-item scales and single-item measures, including five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  All of the scales and single-item measures have a score range from 0 to 100. A high score shows a high response level. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
Quality of Life ELD14 | 36 months
  EORTC QLQ-ELD14 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Module for elderly Cancer patients (14 items), comprising five multi-item and two single-item subscales. The multi-item subscales include questions about mobility (3 items), worries about others (2 items), worries (3 items), maintaining purpose (2 items), and burden of illness (2 items). The single-item subscales include questions related to joint stiffness and Family support. Items are assessed on a 4-level numerical scale with 1= "not at all", 2= "a little", 3= "quite a bit", and 4= "very much". Scores are linearly converted and summated into a scaled score from 0 to 100, with a higher score representing a worse QOL or better QOL for purpose and family support.
Incidence of Treatment-Emergent Adverse Events | 36 months
  AE/SAE evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Ebert, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim, Heidelberg University, II. Medizinische Klinik
Locations (1):
- Universitätsmedizin Mannheim, Heidelberg University, II. Medizinische Klinik, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Meindl-Beinker NM, Maenz M, Betge J, Schulte N, Zhan T, Hofheinz RD, Vogel A, Angermeier S, Bolling C, de Wit M, Jakobs R, Karthaus M, Stocker G, Thuss-Patience P, Leidig T, Bauer H, Ebert MP, Haertel N. Functional status and quality of life in older patients with advanced esophageal squamous cell cancer receiving second-line nivolumab +/- ipilimumab therapy: A post hoc analysis of the phase 2, multicenter RAMONA study. J Geriatr Oncol. 2024 Sep;15(7):101838. doi: 10.1016/j.jgo.2024.101838. Epub 2024 Aug 3. PMID 39097500
- [Derived] Ebert MP, Meindl-Beinker NM, Gutting T, Maenz M, Betge J, Schulte N, Zhan T, Weidner P, Burgermeister E, Hofheinz R, Vogel A, Angermeier S, Bolling C, de Wit M, Jakobs R, Karthaus M, Stocker G, Thuss-Patience P, Leidig T, Gaiser T, Kather JN, Haertel N. Second-line therapy with nivolumab plus ipilimumab for older patients with oesophageal squamous cell cancer (RAMONA): a multicentre, open-label phase 2 trial. Lancet Healthy Longev. 2022 Jun;3(6):e417-e427. doi: 10.1016/S2666-7568(22)00116-7. Epub 2022 Jun 9. PMID 36098320
- [Derived] Meindl-Beinker NM, Betge J, Gutting T, Burgermeister E, Belle S, Zhan T, Schulte N, Maenz M, Ebert MP, Haertel N. A multicenter open-label phase II trial to evaluate nivolumab and ipilimumab for 2nd line therapy in elderly patients with advanced esophageal squamous cell cancer (RAMONA). BMC Cancer. 2019 Mar 14;19(1):231. doi: 10.1186/s12885-019-5446-2. PMID 30871493
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de/
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de/index.html